CLINICAL TRIAL: NCT04220164
Title: Observation of Blood Lipid Outcomes in Patients Who Receive Treatment in Lipid Clinic of Taipei MacKay Memorial Hospital
Brief Title: Observation of Blood Lipid Outcomes in Lipid Clinic
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mackay Memorial Hospital (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 18MMHIS083e
Record Dates: First submitted 2019-12-26; First posted 2020-01-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias | interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dyslipidemic patients: Patients who meet the criteria of high-risk category according to 2017 Taiwan Lipid Guideline for High-Risk Patients have a abnormal serum LDL-C level
  Interventions: Other: Education and inform the optimal threshold of LDL-C levels

INTERVENTIONS:
Other: Education and inform the optimal threshold of LDL-C levels — Physicians educate patients and provide a clear information about optimal LDL-C value according to individual patient's condition according to current guidelines

SUMMARY:
Taipei MacKay Memorial Hospital will establish a Lipid Clinic for hyperlipidemic patients. In this Lipid Clinic, the physician will discuss with each individual patient and set an individualized LDL goal according to current guideline and regulation of National Health Insurance Administration (NHIA). The aim of this study is to observe blood lipid outcomes in patients who receive treatment in Lipid Clinic of Taipei MacKay Memorial Hospital.

DETAILED DESCRIPTION:
Hyperlipidemia is a major risk factor of atherosclerotic cardiovascular disease (ASCVD), and therefore it is beneficial to prevent the risk of ASCVD by controlling the prevalence of hyperlipidemia. According to CEPHEUS Pan-Asia survey, the rate of LDL goal attainment in hyperlipidemic patients of Taiwan was suboptimal, especially in high-risk patients. 2017 Taiwan lipid guideline for high-risk patients has been published and clearly defined the treatment goal of blood LDL-C for high-risk patients. Besides, Taipei MacKay Memorial Hospital will establish a Lipid Clinic for hyperlipidemic patients. In this Lipid Clinic, the physician will discuss with each individual patient and set an individualized LDL goal according to current guideline and regulation of National Health Insurance Administration (NHIA). The aim of this study is to observe blood lipid outcomes in patients who receive treatment in Lipid Clinic of Taipei MacKay Memorial Hospital.

ELIGIBILITY:
Inclusion Criteria:

* ≥20 years-old
* Abnormal lipid profiles according to 2017 Taiwan Lipid Guideline for High-risk Patients

Exclusion Criteria

* Reject to participate in this study
* Pregnant women
* Prisoner
* Illiteracy
* HIV patients
* Individuals who are mentally retarded, homeless, and handicapped

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are ≥20 years, have abnormal lipid profiles, need lipid-lowering drugs according to 2017 Taiwan Lipid Guideline in Lipid Clinic of Taipei MacKay Memorial Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-01-03 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Lipid profile | 12 month
  check serum level of LDL-C

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Feng Lin, PhD, Principal Investigator — Mackay Memorial Hospital
Locations (1):
- Taiwan, Taipei, Mackay Memorial hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
We will not provide IPD to other researchers according to IRB regulation.

REFERENCES:
- [Background] Li YH, Ueng KC, Jeng JS, Charng MJ, Lin TH, Chien KL, Wang CY, Chao TH, Liu PY, Su CH, Chien SC, Liou CW, Tang SC, Lee CC, Yu TY, Chen JW, Wu CC, Yeh HI; Writing Group of 2017 Taiwan Lipid Guidelines for High Risk Patients. 2017 Taiwan lipid guidelines for high risk patients. J Formos Med Assoc. 2017 Apr;116(4):217-248. doi: 10.1016/j.jfma.2016.11.013. Epub 2017 Feb 24. PMID 28242176